CLINICAL TRIAL: NCT05611086
Title: N-Acetylcysteine vs Placebo as Adjunctive Treatment in Pediatric Leukemia: A Single Blind, Randomized Controlled Trial
Brief Title: N-Acetylcysteine vs Placebo as Adjunctive Treatment in Pediatric Leukemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study stopped because the study period already ended
Sponsor: Teny Tjitra Sari (Other)
Responsible Party: Sponsor-Investigator, Teny Tjitra Sari, DR. dr., Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-07-0807
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood
Keywords: Malondialdehyde; N-acetylcysteine; Oxidative stress
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Subjects were randomized consecutively and distributed into two groups. Randomization was done by a third person to decide the distribution of the subjects based on the serial number of randomization.
Who Masked: Participant, Care Provider
Masking Description: Both of the medicines were prepared by the Installation of Pharmacy in Cipto Mangunkusumo National Hospital with the same type and same color of capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC Group (Experimental): Participants of this group was given capsules containing 600mg N-acetylcysteine
  Interventions: Drug: N-Acetylcysteine
- Placebo (Placebo Comparator): Participants of this group was given capsules containing lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — Subjects in treatment group will be given capsules containing 600 mg of NAC
  Other Names: Fluimucil
  Arms: NAC Group
Drug: Placebo — subjects in the control group will be given capsules containing placebo (lactose)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to analyze the effect of N-Acetylcysteine administration towards blood oxidant level, transaminase enzyme, and bilirubin level in ALL children who undergo induction phase of chemotherapy. The main question it aims to answer is whether N-Acetylcysteine can decrease oxidative stress level and reduce hepatotoxicity complication.

Participants will be evaluated for MDA level, transaminase enzymes and bilirubin level before, during, and after the chemotherapy. Participants will be given capsules containing 600mg of N-Acetylcysteine as adjunctive treatment during the 6 weeks induction phase of chemotherapy.

Researchers will compare the lab results to the placebo group to see if there is any significant difference in the results.

DETAILED DESCRIPTION:
The current study has been designed as a randomized single-blind placebo-controlled clinical trial. Sample size calculation for the study was 18 newly diagnosed ALL children in each group using the numerical unpaired two groups data analysis formula. Subjects were recruited from newly diagnosed children with ALL and will start the induction phase of chemotherapy both in hospital ward and outpatient clinic in the Child Health Department at Cipto Mangunkusumo Hospital from August to December 2020. Subjects' parents received an explanation about the study, including the objective and benefits of the study, and also the procedure which will be held. Parents were then asked about the willingness to join the study and signed the form.

Subjects were randomized consecutively and distributed into two groups. Randomization was done by a third person to decide the distribution of the subjects based on the serial number of randomization. Subjects in treatment group will be given capsules containing 600 mg of NAC and subjects in the control group will be given capsules containing placebo (lactose) as the adjunctive treatment during the 6 week induction phase of chemotherapy. Both of the medicines were prepared by the Installation of Pharmacy in Cipto Mangunkusumo National Hospital with the same type and same color of capsules. NAC will be administered during the induction phase of chemotherapy starting in the first week until 6 weeks. This study will analyze change of MDA levels, transaminase enzyme levels, and bilirubin levels before and after the 6th week of the induction phase of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ALL-Standard Risk children who will undergo the induction phase of chemotherapy from 1st week until 6th week
* parents agreed to participate in the study and signed the informed consent

Exclusion Criteria:

* subjects with allergy or contraindicated to consuming N-acetylcysteine
* subjects with liver dysfunction based on clinical and laboratory tests diagnosed before joining the study
* subjects who already consume other antioxidants (vitamin A, vitamin C, and vitamin E).

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
MDA (Malondialdehyde) | Change from Baseline Malondialdehyde level at 7 week
  nanomol
Aspartate aminotransferase | Change from Baseline Aspartate aminotransferase level at 7 week
  u/L
Alanine transaminase | Change from Baseline Alanine transaminase level at 7 week
  u/L
Bilirubin | Change from Baseline Bilirubin level at 7 week
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Teny T Sari, Principal Investigator — DR Cipto Mangunkusumo National Hospital
Locations (1):
- Dr Cipto Mangunkusumo National Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Assessment of the Role of Oxidative Stress and Circulating Biochemical markers in Childhood Leukemia — https://iopscience.iop.org/article/10.1088/1742-6596/1294/6/062089
- See also: Dual effect of oxidative stress on leukemia cancer induction and treatment — https://jeccr.biomedcentral.com/articles/10.1186/s13046-014-0106-5
- See also: Liver Function Tests in Patients of Acute Leukemia before and after Induction Chemotherapy — http://file.scirp.org/html/9-2150920_98373.htm
- See also: Evaluation of Oxidative Stress in Patients with Acute Lymphoblastic Leukemia: Experimental Evidence of the Efficacy of MDA as Cancer Biomarker in Young Patients — http://www.scielo.br/j/jbchs/a/yxBkNvwf7qvTKH9C48zTtcs/abstract/?lang=en